CLINICAL TRIAL: NCT04262882
Title: Development, Testing and Health Effects of a Multilevel Family Planning Intervention
Brief Title: Multilevel Family Planning Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at San Antonio (Other)
Collaborators: Makerere University (Other); San Diego State University (Other); Yale University (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1R21HD098523-01A1 (NIH); 1R21HD098523-01A1 (NIH)
Record Dates: First submitted 2020-02-04; First posted 2020-02-10 (Actual); Results first posted 2023-11-15 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Contraceptive Usage
MeSH Terms: conditions — Contraception Behavior | interventions — Time

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multilevel Family Planning Intervention (Experimental): A multi-level, community-based intervention delivered in groups of couples to increase contraceptive uptake, reduce discontinuation, and reduce the incidence of unintended pregnancy, and improve intermediate outcomes (knowledge, attitudes, norms, communication, equity).
  Interventions: Behavioral: Multilevel Family Planning Intervention
- Time and attention-matched control (Active Comparator): A community sanitation intervention delivered in groups of couples to increase at-home and community hygiene practices.
  Interventions: Behavioral: Time and attention matched control

INTERVENTIONS:
Behavioral: Multilevel Family Planning Intervention — The intervention is comprised of community dialogues, or facilitated discussions, aimed to reshape community norms around gender roles, equity, and family size, and critically analyze the social and community influences of "family-wealth" and poverty with the overall goal of reconstructing individual attitudes and group norms on paths to/definitions of a "successful family" inclusive of family planning. Dialogues are enhanced to address knowledge, motivation, self-efficacy, and relationship dynamics, tailored to men and women. Sessions include both gender segregated and integrated groups with couples in the community.
  Arms: Multilevel Family Planning Intervention
Behavioral: Time and attention matched control — This intervention serves as the attention-matched control. The format and delivery will mirror that of the "Family Health = Family Wealth" intervention (i.e., number, timing, and duration of sessions). The focus of the intervention is on community sanitation and at-home hygiene (hand-washing, food preparation) following an intervention manual that was developed for community groups in Uganda.
  Arms: Time and attention-matched control

SUMMARY:
This study seeks to develop and evaluate a multi-level intervention to satisfy couples' unmet need for family planning in rural Uganda. The study will evaluate the acceptability, feasibility, and preliminary efficacy of the intervention at increasing contraceptive uptake and continuation and improving intermediate outcomes of knowledge, attitudes, perceived community norms, partner communication and equity among couples in rural Uganda.

DETAILED DESCRIPTION:
In 2018, 32.6% of women of reproductive age had an unmet need for family planning in Uganda, meaning they wanted to avoid pregnancy but were not using a modern contraceptive method. Filling the unmet need for family planning has important public health implications, including reductions in pregnancy-related health risks and deaths, and infant mortality. While Uganda is scaling up efforts to reduce supply-side barriers in rural areas, such as community distribution of contraceptives, couples are still faced with multi-level demand-side barriers to contraceptive use. In addition to misinformation and fear of contraceptive side-effects, relationship dynamics, peer and family influence, and broader community norms promoting large family size and traditional gender roles influence family planning. This study will pilot test a multi-level, community-based intervention, which employs transformative community dialogues to alter individual attitudes and the perception of community norms that discourage family planning. Community dialogues are delivered to groups of couples enhanced to simultaneously address individual and interpersonal-level determinants of family planning and link couples to family planning services. The aims of this project are to conduct a pilot quasi-experimental controlled trial to: 1) assess acceptability and feasibility of the trial procedures and intervention content; 2) the intervention's potential efficacy on contraceptive uptake and continuation and intermediate outcomes (knowledge, attitudes, perceived community norms, partner communication and equity) through 6-month follow up.

One village will be randomized to the multi-level intervention and one village to the control condition (attention-matched control intervention). Participation in the full study will last 6 months. Participants will first complete a questionnaire after enrollment, and female participants will take a pregnancy test at baseline. Participants in both study arms will participate in interviewer administered questionnaires at 3 months and 6 months follow-up, pregnancy testing at 6-months follow-up for women, and will permit the research team to access their medical records to extract information about their contraceptive use and use of family planning services. Participants in the intervention arm will participate in a series of group sessions with other couples from the community. Group sessions will last approximately 90 minutes, including community dialogues to reconstruct group norms that discourage contraceptive use enhanced with activities to improve knowledge, motivation, couple dynamics, and link couples to services.

ELIGIBILITY:
Inclusion Criteria:

* Being in a relationship and both partners providing written informed consent; women: age 18-40 (or emancipated minor); men: age 18-50; not currently using modern contraceptives and having never used a non-reversible method; one or both partners wanting to prevent pregnancy for at least the next year; living within the selected villages; Luganda speaking.

Exclusion Criteria:

* Pregnant; Breastfeeding; Using a modern contraceptive method

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2022-05-03 (Actual); Study Completion 2023-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katelyn M Sileo, PhD, MPH, Principal Investigator — University of Texas at San Antonio; Susan M Kiene, PhD, MPH, Principal Investigator — San Diego State University
Locations (2):
- Uganda (2):
  - Katende Villages, Gombe, Butambala
  - Kyabadaza Villages, Gombe, Butambala

IPD SHARING:
Plan to Share IPD: Yes
Quantitative data collected in this trial (baseline, follow-up assessments) will be made available, under the following provisions: (1)The data will be fully de-identified; (2) Access to the data will be made available first to researchers and their students at the four collaborating institutions (within 3 years of study completion): The University of Texas at San Antonio, San Diego State University, the Makerere University School of Public Health (MakSPH), and Yale University; 4) 5 years after study completion, data will be made available to those requesting access outside of the four requesting institutions. Qualitative data collected as part of this trial will not be made available, as it is difficult to fully de-identify and to interpret without knowledge of the context.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 3 years after study completion for researchers and students within the collaborating institutions and 5 years after study completion for those outside of the collaborating institutions upon request
Access Criteria: Upon request from the PI

REFERENCES:
- [Derived] Sileo KM, Muhumuza C, Tuhebwe D, Munoz S, Wanyenze RK, Kershaw TS, Sekamatte S, Lule H, Kiene SM. "The burden is upon your shoulders to feed and take care of your children, not religion or culture": qualitative evaluation of participatory community dialogues to promote family planning's holistic benefits and reshape community norms on family success in rural Uganda. Contracept Reprod Med. 2024 Jun 4;9(1):28. doi: 10.1186/s40834-024-00290-y. PMID 38835058
- [Derived] Sileo KM, Muhumuza C, Sekamatte S, Lule H, Wanyenze RK, Kershaw TS, Kiene SM. The "Family Health = Family Wealth" intervention: study protocol for a pilot quasi-experimental controlled trial of a multi-level, community-based family planning intervention for couples in rural Uganda. Pilot Feasibility Stud. 2022 Dec 24;8(1):265. doi: 10.1186/s40814-022-01226-6. PMID 36564852

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred in May 2021 in 2 communities after they were selected and randomly allocated to either the intervention or comparator arm. Only 2 villages were selected as this was a pilot quasi-experimental controlled trial. Within these two clusters, participants were recruited within couple clusters (units). Recruitment was achieved through household mobilization with support from community health workers who were masked to study purpose and eligibility criteria.
Units Other Than Participants: Couples
Groups:
- Family Health = Family Wealth (FH=FW), Multilevel Family Planning Intervention: FH=FW is a multi-level, community-based intervention delivered in groups of couples to increase contraceptive uptake, reduce discontinuation, and reduce the incidence of unintended pregnancy, and improve intermediate outcomes (knowledge, attitudes, norms, communication, equity).
  FH=FW Intervention: The intervention is comprised of health system strengthening elements paired with community dialogues, or facilitated discussions, aimed to reshape community norms around gender roles, equity, and family size, and critically analyze the social and community influences of "family-wealth" and poverty with the overall goal of reconstructing individual attitudes and group norms on paths to/definitions of a "successful family" inclusive of family planning. Dialogues are enhanced to address knowledge, motivation, self-efficacy, and relationship dynamics, tailored to men and women. Sessions include both gender segregated and integrated groups with couples in the community.
- Time and Attention-matched Comparator Intervention (Water, Sanitation, and Hygiene): A Water, Sanitation, and Hygiene (WASH) intervention delivered in groups of couples to increase at-home and community hygiene practices.
  Time and attention matched control: This intervention serves as the attention-matched comparator intervention. The format and delivery will mirror that of the "Family Health = Family Wealth" intervention (i.e., number, timing, and duration of sessions). The focus of the intervention is on community sanitation and at-home hygiene (hand-washing, food preparation) following an intervention manual that was developed for community groups in Uganda.
Period: Overall Study
Arm/Group | Family Health = Family Wealth (FH=FW), Multilevel Family Planning Intervention | Time and Attention-matched Comparator Intervention (Water, Sanitation, and Hygiene)
Started | 84; 42 Couples | 76; 38 Couples
Completed | 69; 35 Couples | 70; 35 Couples
Not Completed | 15; 7 Couples | 6; 3 Couples
Not completed — Investigator withdrawal due to non-attendance of session 1 (at least 1 person in couple) | 14 | 6
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: The baseline sample excludes the participants withdrawn and replaced by investigators, considered the final sample of 140 individuals, or 70 couples. Individual participants are nested within couples. The unit of analysis, however, for all baseline data presented is the individual, as all demographic measures were collected from individuals.
Units Other Than Participants: Couples
Groups:
- Total: Total of all reporting groups
Arm/Group | Family Health = Family Wealth (FH=FW), Multilevel Family Planning Intervention | Time and Attention-matched Comparator Intervention (Water, Sanitation, and Hygiene) | Total
Number analyzed (Participants) | 70 | 70 | 140
Number analyzed (Couples) | 35 | 35 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.01 (6.79) | 30.77 (8.27) | 29.89 (7.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 35 | 70
  Male | 35 | 35 | 70
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 70 | 70 | 140
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Religion [Count of Participants; unit: Participants]
  Catholic, Protestant, and Other | 36 | 22 | 58
  Muslim | 34 | 48 | 82

OUTCOME MEASURES:

1. Primary Outcome: Number of Couples With Uptake of Any High Efficacy Contraceptive Method
Description: Uptake of any high efficacy contraceptive method. High efficacy contraceptive methods are defined based on efficacy for "typical use" of methods (rather than perfect use), inclusive of pills, injection, intrauterine device, implant, tubal ligation, vasectomy; measured through women's self-report and validated through clinic records and men's self-report
Time Frame: 7-months and 10-months follow-up
Population: Couple is the unit of analysis; one outcome per couple
Measure: Count of Units; unit: Couple
Units Other Than Participants: Couple
Arm/Group | Family Health = Family Wealth (FH=FW), Multilevel Family Planning Intervention | Time and Attention-matched Comparator Intervention (Water, Sanitation, and Hygiene)
Number analyzed (Participants) | 69 | 70
Number analyzed (Couple) | 35 | 35
Couple
  7-months: Yes, using method | 20 | 9
  7-months: No, not using method | 15 | 26
  10-months: Yes, using method | 20 | 6
  10-months: No, not using method | 15 | 29
Statistical Analysis 1: Comparison: Family Health = Family Wealth (FH=FW), Multilevel Family Planning Intervention vs Time and Attention-matched Comparator Intervention (Water, Sanitation, and Hygiene); Test type: Superiority; p = 0.20, Regression, Logistic; Adjusted for age and religion. Analysis in GEE to account for dependence in repeated, dyadic data; Odds Ratio (OR) = 1.67, 95% CI 2-sided [0.77 to 3.64] — Reference group is the comparator arm

2. Secondary Outcome: Number of Couples That Discontinued Use of a High Efficacy Contraceptive Method at 10-months Follow-up Among Those That Started Using a Method at 7-months Follow-up
Description: Number of couples that discontinued use of a high efficacy contraceptive method at 10-months follow-up among those that started using a method at 7-months follow-up. High efficacy contraceptive methods are defined based on efficacy for "typical use" of methods (rather than perfect use), inclusive of pills, injection, intrauterine device, implant, tubal ligation, vasectomy; measured through women's self-report and validated through clinic records and men's self-report
Time Frame: 7 and 10 months follow-up
Population: Number analyzes includes participants that began using a high efficacy contraceptive method at 7-months follow-up
Measure: Count of Units; unit: Couples
Units Other Than Participants: Couples
Arm/Group | Family Health = Family Wealth (FH=FW), Multilevel Family Planning Intervention | Time and Attention-matched Comparator Intervention (Water, Sanitation, and Hygiene)
Number analyzed (Participants) | 40 | 18
Number analyzed (Couples) | 20 | 9
Couples | 2 | 3

3. Secondary Outcome: Number of Couples With an Unintended Pregnancy
Description: Biological measure; human chorionic gonadotropin (hCG) rapid pregnancy tests taken by women at 10-months follow-up.
Time Frame: 10-months follow-up
Population: Couple is the unit of analysis (one outcome per couple)
Measure: Count of Units; unit: Couple
Units Other Than Participants: Couple
Arm/Group | Family Health = Family Wealth (FH=FW), Multilevel Family Planning Intervention | Time and Attention-matched Comparator Intervention (Water, Sanitation, and Hygiene)
Number analyzed (Participants) | 69 | 70
Number analyzed (Couple) | 35 | 35
Couple
  Yes, unintended pregnancy | 1 | 1
  No unintended pregnancy | 34 | 34

4. Secondary Outcome: Change in Knowledge of Contraceptives
Description: Scale from the Uganda Demographic and Health Survey (DHS) aimed to assess knowledge of modern contraceptive methods; collected through interviewer-administered questionnaire. Possible range 0-1, greater scores indicate more knowledge
Time Frame: Baseline, 7 and 10 months follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Family Health = Family Wealth (FH=FW), Multilevel Family Planning Intervention | Time and Attention-matched Comparator Intervention (Water, Sanitation, and Hygiene)
Number analyzed (Participants) | 69 | 70
score on a scale
  Baseline | 0.63 (0.32) | 0.52 (0.22)
  7-months | 0.99 (0.26) | 0.62 (0.15)
  10-months | 1.00 (0.00) | 0.59 (0.16)
Statistical Analysis 1: Comparison: Family Health = Family Wealth (FH=FW), Multilevel Family Planning Intervention vs Time and Attention-matched Comparator Intervention (Water, Sanitation, and Hygiene); Test type: Superiority; p < 0.001, Regression, Linear; Models control for age and religion. Models run using generalized estimating equations (GEE) to account for dependence in repeated, dyadic data; Wald Chi-Square = 35.20 — Wald Chi-Square tests the overall arm*time intervention effect across the timepoints
Statistical Analysis 2: Comparison: Family Health = Family Wealth (FH=FW), Multilevel Family Planning Intervention vs Time and Attention-matched Comparator Intervention (Water, Sanitation, and Hygiene); Test type: Superiority; p < 0.001, Regression, Linear — P-value is adjusted for multiple comparisons; this value is for the 7-month follow-up; [statistical method as in outcome 4, analysis 1]; unstandardized beta = 0.41, Standard Error of Mean 0.07
Statistical Analysis 3: Comparison: Family Health = Family Wealth (FH=FW), Multilevel Family Planning Intervention vs Time and Attention-matched Comparator Intervention (Water, Sanitation, and Hygiene); Test type: Superiority; p < 0.001, Regression, Linear — P-value is adjusted for multiple comparisons; this value is for the 10-month follow-up; [statistical method as in outcome 4, analysis 1]; unstandardized beta = 0.40, Standard Error of Mean 0.07

5. Secondary Outcome: Change in Family Planning Attitudes
Description: Family planning attitudes scale developed for use in Uganda to assess how participants would feel about using contraceptive methods; collected through interviewer-administered questionnaire. Scores range from 0-4 with greater scores indicating more positive attitudes towards family planning.
Time Frame: Baseline, 7 and 10 months follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Family Health = Family Wealth (FH=FW), Multilevel Family Planning Intervention | Time and Attention-matched Comparator Intervention (Water, Sanitation, and Hygiene)
Number analyzed (Participants) | 69 | 70
score on a scale
  Baseline | 2.76 (0.51) | 2.58 (0.55)
  7-months | 3.56 (0.39) | 2.23 (0.62)
  10-months | 3.27 (0.32) | 2.22 (0.57)
Statistical Analysis 1: Comparison: Family Health = Family Wealth (FH=FW), Multilevel Family Planning Intervention vs Time and Attention-matched Comparator Intervention (Water, Sanitation, and Hygiene); Test type: Superiority; p < 0.001, Regression, Linear — Models control for age and religion. Models run using generalized estimating equations (GEE) to account for dependence in repeated, dyadic data; Wald Chi-Square = 64.53 — Wald Chi-Square tests the overall arm*time intervention effect across the timepoints; Tests of significance for each follow-up time point: 7-months: unstandardized beta=1.08, standard error=0.14, p < 0.001; 10-months: unstandardized beta=0.79, standard error=0.14, p < 0.001
Statistical Analysis 2: Comparison: Family Health = Family Wealth (FH=FW), Multilevel Family Planning Intervention vs Time and Attention-matched Comparator Intervention (Water, Sanitation, and Hygiene); Test type: Superiority; p < 0.001, Regression, Linear — Adjusted for multiple comparisons; this value is for the 7-month follow-up; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = 1.08, Standard Error of Mean 0.14
Statistical Analysis 3: Comparison: Family Health = Family Wealth (FH=FW), Multilevel Family Planning Intervention vs Time and Attention-matched Comparator Intervention (Water, Sanitation, and Hygiene); Test type: Superiority; p < 0.001, Regression, Linear — Adjusted for multiple comparisons; this value is for the 10-month follow-up; [statistical method as in outcome 4, analysis 1]; unstandardized beta = 0.79, Standard Error of Mean 0.14

6. Secondary Outcome: Change in Perceived Family Planning Norms
Description: Scale adapted from the Family Planning Approval Index to assess the perceived acceptance of family planning and contraceptive use among partner, family, peers, and broader community; collected through interviewer-administered questionnaire. Scores range from 0-1 with greater scores indicating more positive perceived attitudes towards family planning among others
Time Frame: Baseline, 7 and 10 months follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Family Health = Family Wealth (FH=FW), Multilevel Family Planning Intervention | Time and Attention-matched Comparator Intervention (Water, Sanitation, and Hygiene)
Number analyzed (Participants) | 69 | 70
score on a scale
  Baseline | 0.86 (0.21) | 0.93 (0.21)
  7-months | 0.96 (0.12) | 0.75 (0.36)
  10-months | 0.95 (0.13) | 0.87 (0.28)
Statistical Analysis 1: Comparison: Family Health = Family Wealth (FH=FW), Multilevel Family Planning Intervention vs Time and Attention-matched Comparator Intervention (Water, Sanitation, and Hygiene); Test type: Superiority; p < 0.001, Regression, Linear; [statistical method as in outcome 4, analysis 1]; Wald Chi-Square = 23.89
Statistical Analysis 2: Comparison: Family Health = Family Wealth (FH=FW), Multilevel Family Planning Intervention vs Time and Attention-matched Comparator Intervention (Water, Sanitation, and Hygiene); Test type: Superiority; p < 0.001, Regression, Linear — P value is adjusted for multiple comparisons; this value is for the 7-month follow-up; [statistical method as in outcome 4, analysis 1]; unstandardized beta = 0.31, Standard Error of Mean 0.06
Statistical Analysis 3: Comparison: Family Health = Family Wealth (FH=FW), Multilevel Family Planning Intervention vs Time and Attention-matched Comparator Intervention (Water, Sanitation, and Hygiene); Test type: Superiority; p < 0.001, Regression, Linear — P-value is adjusted for multiple comparisons; this value is for the 10-month follow-up; [statistical method as in outcome 4, analysis 1]; unstandardized beta = 0.19, Standard Error of Mean 0.05

7. Secondary Outcome: Change in Family Planning Intentions
Description: Family planning intentions scale developed for use in Uganda to assess participants' plans to use contraceptives and family planning services in the future; collected through interviewer-administered questionnaire. Scores range between 0-4 with higher scores indicating greater intentions to use family planning services in the future
Time Frame: Baseline, 7 and 10 months follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Family Health = Family Wealth (FH=FW), Multilevel Family Planning Intervention | Time and Attention-matched Comparator Intervention (Water, Sanitation, and Hygiene)
Number analyzed (Participants) | 69 | 70
score on a scale
  Baseline | 3.14 (0.43) | 2.20 (0.59)
  7-montha | 3.65 (0.42) | 2.02 (0.97)
  10 months | 3.22 (0.36) | 2.12 (0.63)
Statistical Analysis 1: Comparison: Family Health = Family Wealth (FH=FW), Multilevel Family Planning Intervention vs Time and Attention-matched Comparator Intervention (Water, Sanitation, and Hygiene); Test type: Superiority; p < 0.001, Regression, Linear; Models control for age and religion. Models were run using generalized estimating equations (GEE) to account for dependence in repeated, dyadic data; Wald Chi-Square = 48.26
Statistical Analysis 2: Comparison: Family Health = Family Wealth (FH=FW), Multilevel Family Planning Intervention vs Time and Attention-matched Comparator Intervention (Water, Sanitation, and Hygiene); Test type: Superiority; p < 0.001, Regression, Cox — P-value is adjusted for multiple comparisons; this value is for the 7-month follow-up; [statistical method as in outcome 4, analysis 1]; unstandardized beta = 0.68, Standard Error of Mean 0.12
Statistical Analysis 3: Comparison: Family Health = Family Wealth (FH=FW), Multilevel Family Planning Intervention vs Time and Attention-matched Comparator Intervention (Water, Sanitation, and Hygiene); Test type: Superiority; p = 0.04, Regression, Linear — P-value is adjusted for multiple comparisons; this value is for the 10-month follow-up; [statistical method as in outcome 4, analysis 1]; unstandardized beta = 0.20, Standard Error of Mean 0.10

8. Secondary Outcome: Change in Desired Number of Children (Fertility Desires)
Description: Item from the Uganda Demographic and Health Survey (DHS) on the participants' fertility desires (i.e., desired number of additional children); collected through interviewer-administered questionnaire. This is a count variable that could range from zero upward (no limit).
Time Frame: Baseline, 7 and 10 months follow-up
Measure: Mean (Standard Deviation); unit: desired additional children
Arm/Group | Family Health = Family Wealth (FH=FW), Multilevel Family Planning Intervention | Time and Attention-matched Comparator Intervention (Water, Sanitation, and Hygiene)
Number analyzed (Participants) | 69 | 70
desired additional children
  Baseline | 2.90 (1.49) | 2.76 (2.59)
  7-months | 2.38 (1.24) | 2.47 (1.40)
  10-months | 1.83 (0.64) | 2.36 (1.38)
Statistical Analysis 1: Comparison: Family Health = Family Wealth (FH=FW), Multilevel Family Planning Intervention vs Time and Attention-matched Comparator Intervention (Water, Sanitation, and Hygiene); Test type: Superiority; p = 0.007, Regression, Linear — Arm*Time p value for 10-months follow up overall; Model controls for age and religion. Model was run using generalized estimating equations (GEE) to account for dependence in repeated, dyadic data; Wald Chi-Square = 9.87
Statistical Analysis 2: Comparison: Family Health = Family Wealth (FH=FW), Multilevel Family Planning Intervention vs Time and Attention-matched Comparator Intervention (Water, Sanitation, and Hygiene); Test type: Superiority — Models control for age and religion. Models run using generalized estimating equations (GEE) to account for dependence in repeated, dyadic data; p = 0.60, Regression, Linear — P-value is adjusted for multiple comparisons; this value is for the 7-month follow-up; unstandardized beta = -0.16, Standard Error of Mean 0.32
Statistical Analysis 3: Comparison: Family Health = Family Wealth (FH=FW), Multilevel Family Planning Intervention vs Time and Attention-matched Comparator Intervention (Water, Sanitation, and Hygiene); Test type: Superiority; p = 0.07, Regression, Linear — P-value is adjusted for multiple comparisons; this value is for the 10-month follow-up; [statistical method as in outcome 4, analysis 1]; Slope = -0.53, Standard Error of Mean 0.07

9. Secondary Outcome: Change in Fertility Discordance Between Partners
Description: An item from the Uganda DHS on the participants' desired number of children, "How many more children do you want to have?" was used to calculate the couple variable fertility discordance by subtracting men and women's responses within couples. This was dichotomized for analysis; for couples where the product was zero, they were classified as having no discordance (0) and for couples where the produce was anything other than zero, they were classified as having discordance (1).
Time Frame: Baseline, 7 and 10 months follow-up
Measure: Count of Units; unit: Couples
Units Other Than Participants: Couples
Arm/Group | Family Health = Family Wealth (FH=FW), Multilevel Family Planning Intervention | Time and Attention-matched Comparator Intervention (Water, Sanitation, and Hygiene)
Number analyzed (Participants) | 69 | 70
Number analyzed (Couples) | 35 | 35
Couples
  Baseline | 15 | 18
  7-months | 19 | 12
  10-months | 3 | 27
Statistical Analysis 1: Comparison: Family Health = Family Wealth (FH=FW), Multilevel Family Planning Intervention vs Time and Attention-matched Comparator Intervention (Water, Sanitation, and Hygiene); Test type: Superiority; p = 0.005, Regression, Logistic; [statistical method as in outcome 8, analysis 1]; Wald Chi-Square = 10.42
Statistical Analysis 2: Comparison: Family Health = Family Wealth (FH=FW), Multilevel Family Planning Intervention vs Time and Attention-matched Comparator Intervention (Water, Sanitation, and Hygiene); Test type: Superiority; p = 0.05, Regression, Logistic — P-value is adjusted for multiple comparisons; this value is for the 7-month follow-up; [statistical method as in outcome 4, analysis 1]; Odds Ratio (OR) = 1.36, 95% CI 2-sided [0.99 to 1.85]
Statistical Analysis 3: Comparison: Family Health = Family Wealth (FH=FW), Multilevel Family Planning Intervention vs Time and Attention-matched Comparator Intervention (Water, Sanitation, and Hygiene); Test type: Superiority; p = 0.71, Regression, Logistic — P-value is adjusted for multiple comparisons; this value is for the 10-month follow-up; [statistical method as in outcome 4, analysis 1]; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.75 to 1.22]

10. Secondary Outcome: Change in Joint Household Decision-making
Description: Joint household decision-making was measured with four items from the Uganda DHS that ask respondents who primarily decides on: 1) how the money they earn is used; 2) how their spouses' earnings are used; 3) decisions about healthcare for yourself; and 4) decisions about major household purchases. Response options were recoded as self and partner jointly (1) vs. all other (0). A mean score was calculated for each time point with greater scores indicating more joint decision-making (range 0-1).
Time Frame: Baseline, 7 and 10 months follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Family Health = Family Wealth (FH=FW), Multilevel Family Planning Intervention | Time and Attention-matched Comparator Intervention (Water, Sanitation, and Hygiene)
Number analyzed (Participants) | 69 | 70
score on a scale
  Baseline | 0.75 (0.29) | 0.84 (0.26)
  7-months | 0.97 (0.17) | 0.91 (0.23)
  10-months | 1.00 (0.00) | 0.87 (0.19)
Statistical Analysis 1: Comparison: Family Health = Family Wealth (FH=FW), Multilevel Family Planning Intervention vs Time and Attention-matched Comparator Intervention (Water, Sanitation, and Hygiene); Test type: Superiority; p = 0.001, Regression, Linear; [statistical method as in outcome 8, analysis 1]; Wald Chi-Square = 13.40
Statistical Analysis 2: Comparison: Family Health = Family Wealth (FH=FW), Multilevel Family Planning Intervention vs Time and Attention-matched Comparator Intervention (Water, Sanitation, and Hygiene); Test type: Superiority; p = 0.07, Regression, Linear — P-value is adjusted for multiple comparisons; this value is for the 7-month follow-up; [statistical method as in outcome 4, analysis 1]; unstandardized beta = 0.13, Standard Error of Mean 0.07
Statistical Analysis 3: Comparison: Family Health = Family Wealth (FH=FW), Multilevel Family Planning Intervention vs Time and Attention-matched Comparator Intervention (Water, Sanitation, and Hygiene); Test type: Superiority; p < 0.001, Regression, Linear — P-value is adjusted for multiple comparisons; this value is for the 10-month follow-up; [statistical method as in outcome 4, analysis 1]; unstandardized beta = 0.21, Standard Error of Mean 0.06

11. Secondary Outcome: Change in Partner Communication About Family Planning
Description: The mean of two items on the frequency of communication with one's partner about family planning found predictive of family planning in Uganda in prior research. Participants were asked, in the last 12 months, "How often have you discussed the number of children you want with your partner?" and "How often have you discussed the spacing or timing of your/your partner's pregnancies with your partner." The four-point response options ranged from "Never" to "Regularly." At the two follow-up time points, the same questions were asked with the timeframe, "since the last interview." Higher scores indicate more communication. Possible scores range from 0.00-3.00.
Time Frame: Baseline, 7 and 10 months follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Family Health = Family Wealth (FH=FW), Multilevel Family Planning Intervention | Time and Attention-matched Comparator Intervention (Water, Sanitation, and Hygiene)
Number analyzed (Participants) | 69 | 70
score on a scale
  Baseline | 1.89 (0.73) | 1.82 (0.46)
  7-months | 2.84 (0.34) | 1.61 (0.54)
  10-months | 2.61 (0.48) | 0.91 (0.70)
Statistical Analysis 1: Comparison: Family Health = Family Wealth (FH=FW), Multilevel Family Planning Intervention vs Time and Attention-matched Comparator Intervention (Water, Sanitation, and Hygiene); Test type: Superiority; p = 0.001, Regression, Linear; [statistical method as in outcome 8, analysis 1]; Wald Chi-Square = 78.81
Statistical Analysis 2: Comparison: Family Health = Family Wealth (FH=FW), Multilevel Family Planning Intervention vs Time and Attention-matched Comparator Intervention (Water, Sanitation, and Hygiene); Test type: Superiority; p < 0.001, Regression, Linear — P-value is adjusted for multiple comparisons; this value is for the 7-month follow-up; [statistical method as in outcome 4, analysis 1]; unstandardized beta = 1.19, Standard Error of Mean 0.18
Statistical Analysis 3: Comparison: Family Health = Family Wealth (FH=FW), Multilevel Family Planning Intervention vs Time and Attention-matched Comparator Intervention (Water, Sanitation, and Hygiene); Test type: Superiority; p = 0.001, Regression, Linear — P-value is adjusted for multiple comparisons; this value is for the 10-month follow-up; [statistical method as in outcome 4, analysis 1]; unstandardized beta = 1.65, Standard Error of Mean 0.19

12. Secondary Outcome: Change in Gender Inequitable Attitudes
Description: The mean of the 24-item Gender Equitable Men scale measured endorsement of traditional gender norms and attitudes on gender inequity, validated in Tanzania and Ghana, with good reliability in African settings. Domains include violence, sexual relationships, reproductive health and disease prevention, and domestic chores and daily life items. Higher scores indicate more inequitable gender attitudes. Possible score range = 0=3
Time Frame: Baseline, 7 and 10 months follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Family Health = Family Wealth (FH=FW), Multilevel Family Planning Intervention | Time and Attention-matched Comparator Intervention (Water, Sanitation, and Hygiene)
Number analyzed (Participants) | 69 | 70
score on a scale
  Baseline | 1.41 (0.24) | 1.70 (0.20)
  7-months | 1.32 (0.18) | 1.74 (0.12)
  10-months | 1.33 (0.12) | 1.80 (0.09)
Statistical Analysis 1: Comparison: Family Health = Family Wealth (FH=FW), Multilevel Family Planning Intervention vs Time and Attention-matched Comparator Intervention (Water, Sanitation, and Hygiene); Test type: Superiority; p < 0.001, Regression, Linear; [statistical method as in outcome 8, analysis 1]; Wald Chi-Square = 19.46
Statistical Analysis 2: Comparison: Family Health = Family Wealth (FH=FW), Multilevel Family Planning Intervention vs Time and Attention-matched Comparator Intervention (Water, Sanitation, and Hygiene); Test type: Superiority; p = 0.008, Regression, Linear — P-value is adjusted for multiple comparisons; this value is for the 7-month follow-up; [statistical method as in outcome 4, analysis 1]; unstandardized beta = -0.13, Standard Error of Mean 0.05
Statistical Analysis 3: Comparison: Family Health = Family Wealth (FH=FW), Multilevel Family Planning Intervention vs Time and Attention-matched Comparator Intervention (Water, Sanitation, and Hygiene); Test type: Superiority; p < 0.001, Regression, Linear — P-value is adjusted for multiple comparisons; this value is for the 10-month follow-up; [statistical method as in outcome 4, analysis 1]; unstandardized beta = -0.17, Standard Error of Mean 0.04

ADVERSE EVENTS:
Time Frame: 10 months
Arm/Group | Family Health = Family Wealth (FH=FW), Multilevel Family Planning Intervention | Time and Attention-matched Comparator Intervention (Water, Sanitation, and Hygiene)
All-Cause Mortality (participants affected / at risk) | 0/84 | 0/76
Serious Adverse Events (participants affected / at risk) | 0/84 | 0/76
Other Adverse Events (participants affected / at risk) | 0/84 | 0/76

LIMITATIONS AND CAVEATS:
This was a pilot quasi-experimental controlled trial with the primary aims of establishing acceptability, feasibility, and preliminary effects of the intervention on the main and secondary outcomes. Thus, the intervention needs to be tested in a fully powered cluster randomized controlled trial to establish intervention efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-16): https://cdn.clinicaltrials.gov/large-docs/82/NCT04262882/Prot_SAP_000.pdf